CLINICAL TRIAL: NCT00761345
Title: Phase I Study of Low-Dose Fractionated Radiotherapy as a Chemosensitizer for Gemcitabine and Erlotinib in Patients With Locally Advanced or Limited Metastatic Pancreatic Cancer
Brief Title: Study of Low-Dose Fractionated Radiotherapy in Patients With Locally Advanced Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-GI-021; OSI4485s (Other: Genentech)
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Pancreatic Carcinoma Non-resectable; Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; locally advanced; unresectable; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy and chemotherapy (Experimental): gemcitabine will be administered at 1000mg/m2 IV on days 1 and 8 of each 21 day cycle. erlotinib at either 100mg (cohort 1-3) or 150mg (cohort 4) PO daily. Low dose fractionated radiotherapy (LDRT) will be given BID on days 1 and 2 and 8 and 9 of each 21 day cycle
  Interventions: Drug: gemcitabine; Drug: Erlotinib; Radiation: low dose fractionated radiotherapy

INTERVENTIONS:
Drug: gemcitabine — gemcitabine 1000mg/m2 days 1 and 8 of each 21 day cycle.
  Other Names: Gemzar
Drug: Erlotinib — Erlotinib 100mg or 150mg daily of each 21 day cycle
  Other Names: Tarceva
Radiation: low dose fractionated radiotherapy — low dose fractionated radiotherapy day 1 and 2, day 8 and 9 of each 21 day cycle

SUMMARY:
People with pancreatic cancer usually have a large amount of the cancer in the area of the pancreas and around it when they are diagnosed with it. Or their cancer has spread (metastasized)outside that area of the abdomen and is not able to be surgically removed (resected). For patients with metastatic disease, one standard treatment is the combination of gemcitabine and erlotinib. This combination has shown slightly longer survival compared to getting gemcitabine alone. For patients with localized but unresectable disease, the standard treatment remains controversial. Early studies showed that chemotherapy and radiation together was better than either one used alone. The greatest benefit of external beam radiotherapy may be after a period of full-dose chemotherapy alone, to help the rapid spread. A problem of beginning treatment with standard radiotherapy is that the doses of chemotherapy usually have to be reduced sometimes by half.

Studies have already shown that low dose radiotherapy (LDRT)is safe. This study will evaluate the safety of LDRT instead of standard doses with full dosing of gemcitabine and erlotinib in patients with locally advanced or limited metastatic pancreatic cancer. Patients will be enrolled in groups of 3 to 6 each with a slightly higher dose of LDRT and erlotinib.

For patients with locally advanced disease, this protocol also may help because most patients develop and die from spread to the liver and abdominal cavity.

DETAILED DESCRIPTION:
Pancreatic cancer is nearly universally fatal, with approximately 38,000 new cases and 34,000 deaths expected in 2008.1 The majority of patients present with disease that is not amenable to curative resection. For patients with metastatic disease, one standard treatment is the combination of gemcitabine with the small molecule epidermal growth factor tyrosine kinase inhibitor erlotinib. This combination results in a modest survival benefit compared to single agent gemcitabine.2

For patients presenting with localized but unresectable disease, the standard treatment remains controversial. Early studies demonstrated that chemotherapy and radiation was superior to either modality alone.3 However, recent studies of systemic therapy alone have typically included a small but real minority of patients with locally advanced disease, supporting that systemic therapy alone is a reasonable treatment option.2 Adding to the confusion are recent European reports that systemic therapy alone may be superior to combined modality therapy, at least when used initially.4 The greatest benefit of external beam radiotherapy may be after a period of full-dose chemotherapy alone, to ensure that rapid metastases do not develop.5 A limitation of beginning treatment with conventional external beam radiotherapy is a requirement to reduce dosing of gemcitabine by 40-50%. Given the safety and preclinical rationale for LDRT, we propose this phase I study to evaluate the safety of LDRT with standard dosing of gemcitabine and erlotinib in patients with locally advanced or limited metastatic pancreatic cancer. Patients will be enrolled in cohorts with escalating doses of low dose radiotherapy. Radiation ports will be uniform between patients as described in Section 5.6 below. As LDRT is administered to sites of disease in liver and abdominal cavity to iliac crest, patients with metastatic disease confined to these areas will be eligible. For patients with locally advanced disease, this protocol also has high rationale, as the overwhelming majority of patients develop and succumb to recurrences in liver and abdominal cavity,10 areas which would be covered by the proposed radiation field. The dose of 2880 cGy is the limit because of kidney and other upper abdominal organ potential for toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of adenocarcinoma of the pancreas that is not amenable to curative surgical resection. Patients with locally advanced unresectable disease and those patients with metastatic disease that can be encompassed in the radiation fields for this study (as assessed by treating radiation oncologist) are eligible.
* Patients may not have received any prior chemotherapy for locally advanced or metastatic pancreatic cancer. Prior adjuvant chemotherapy completed >1 year previously is allowed.
* Patients must be able to provide informed consent and HIPAA consent.
* Patients must be ≥18 years of age
* Adequate hematologic and organ function:

  * ANC ≥ 1,000/μL, platelets ≥ 100,000/μL, hemoglobin ≥ 9.0/dL
  * Bilirubin: ≤1.5X ULN
  * ALT/AST < 3.0 X upper limit of normal
  * Serum Creatinine: WNL
  * Albumin > 2.5 g/dL
* Measurable and non-measurable disease are permitted
* ECOG performance status 0-1
* Patients must be able to swallow oral medications
* Patients must be able to comply with study and follow up procedures

Exclusion Criteria:

* No prior radiation therapy to the abdomen.
* Patients must not have any other active illness (e.g. active/uncontrolled infection, uncontrolled cardiac disease, etc.) that would preclude safe therapy in the judgment of the treating physicians. Patients may be enrolled while still on antibiotics as long as clinical signs of active infection are absent.
* Patients with concurrent active malignancy requiring therapy are not eligible. Patients with a history of malignancy within any timeframe not requiring ongoing therapy are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Karmanos Cancer Institue, Detroit, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Reading Medical Center, West Reading, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiotherapy and Chemotherapy
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Patients with locally advanced or metastatic pancreatic cancer confined to the abdomen and an ECOG performance status (PS) of 0-1 who had received 0-1 prior regimens (without Gemcitabine or Erlotinib) and no prior radiotherapy were eligible
Arm/Group | Radiotherapy and Chemotherapy
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Dose Limiting Toxicities
Time Frame: weekly physician and nurse assessment and in between as needed until 30 days after treatment termination
Population: 27 patients (median age 64years and 15 male) with locally advanced or metastatic pancreatic cancer confined to the abdomen and an ECOG performance status of 0-1 who had received 0-1 prior regimens (without Gemcitabine or Erlotinib) and no prior radiotherapy were eligible.
Measure: Number; unit: participants
Arm/Group | Radiotherapy and Chemotherapy
Number analyzed (Participants) | 27
participants | 27

2. Secondary Outcome: To Measure Progression Free Survival and Overall Survival
Time Frame: Evaluate CT scans after every 2 cycles of therapy (about every 6 weeks) and long term follow up every 3 months once off treatment for survival
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3.5 years
Arm/Group | Radiotherapy and Chemotherapy
Serious Adverse Events (participants affected / at risk) | 15/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy and Chemotherapy (N=27)
Ileus (Gastrointestinal disorders) | 2 (2)
DVT (Vascular disorders) | 2 (2)
GI bleed (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Biliary obstruction (Hepatobiliary disorders) | 1 (1)
Perforated viscous (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy and Chemotherapy (N=27)
hemoglobin (Blood and lymphatic system disorders) | 25 (120)
ANC (Blood and lymphatic system disorders) | 14 (41)
WBC (Blood and lymphatic system disorders) | 22 (84)
Platelets (Blood and lymphatic system disorders) | 19 (68)
Edema (General disorders) | 6 (15)
DVT (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (3)
Fever (General disorders) | 6 (13)
Fatigue (General disorders) | 26 (107)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (5)
watery eyes (Eye disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 18 (61)
Dry desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Dry cracked skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Jaundice (Hepatobiliary disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (18)
GI bleed (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (53)
Vomiting (Gastrointestinal disorders) | 13 (35)
Dysphagia (Gastrointestinal disorders) | 4 (6)
Dyspesia (Gastrointestinal disorders) | 5 (10)
Heartburn (Gastrointestinal disorders) | 3 (12)
Constipation (Gastrointestinal disorders) | 10 (27)
Ileus/bowel obstruction (Gastrointestinal disorders) | 1 (1)
Bowel perforation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 22 (65)
Dehydration (Metabolism and nutrition disorders) | 8 (14)
Mucositis (Gastrointestinal disorders) | 1 (2)
Dysgeusia (Gastrointestinal disorders) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 21 (69)
Hemorrhoids (Gastrointestinal disorders) | 1 (3)
Weight loss (Metabolism and nutrition disorders) | 14 (43)
Insomnia (Psychiatric disorders) | 7 (15)
Depression (Psychiatric disorders) | 10 (32)
Neuropathy, sensory (Nervous system disorders) | 1 (5)
Tremor (Nervous system disorders) | 2 (8)
Pain (General disorders) | 16 (47)
Abdominal pain (Gastrointestinal disorders) | 12 (32)
Headache (Nervous system disorders) | 1 (1)
Myalgia/Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (19)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 5 (6)
Alkaline phosphatase (Investigations) | 15 (51)
Creatinine (Investigations) | 7 (10)
SGOT/AST (Investigations) | 12 (18)
SGPT/ALT (Investigations) | 7 (10)
Infection, without neurtropenia (Infections and infestations) | 6 (10)
Infection, with neutropenia (Infections and infestations) | 1 (1)
Hyperglycemia (Investigations) | 18 (60)
Hypoglycemia (Investigations) | 2 (2)
Hypoalbuminemia (Investigations) | 23 (94)
Hypokalemia (Investigations) | 16 (38)
Hyponatremia (Investigations) | 16 (35)
Hypocalcemia (Investigations) | 8 (17)
Lymphopenia (Investigations) | 7 (19)
Hypomagnesemia (Investigations) | 6 (9)
Low bicarbonate (Investigations) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Radiation dermititis (Skin and subcutaneous tissue disorders) | 1 (3)
Tachycardia (Cardiac disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Chills (General disorders) | 1 (2)
Sweats (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes